CLINICAL TRIAL: NCT03268421
Title: Multi-site Randomized Clinical Trial of FIT Teens for Juvenile Fibromyalgia
Brief Title: Fibromyalgia Integrative Training for Adolescents With Juvenile Fibromyalgia
Acronym: FIT Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIN001-FIT Teens; R01AR070474 (NIH)
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia; Myofascial Pain Syndrome; Muscular Diseases; Musculoskeletal Disease; Rheumatic Diseases
Keywords: juvenile fibromyalgia; pain in children; musculoskeletal pain; cognitive behavioral therapy; coping skills training; neuromuscular exercise; graded aerobic exercise
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes; Muscular Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Musculoskeletal Pain | interventions — Cognitive Behavioral Therapy; Coping Skills

STUDY DESIGN:
Intervention Model Description: Non-pharmacologic trial comparing behavioral and exercise-based treatments
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fibromyalgia Integrative Training for Teens (Experimental): Fibromyalgia Integrative Training for Teens (FIT Teens) is a combined coping skills training and physical exercise program. Pain coping skills training, also called cognitive behavioral therapy (CBT) teaches a number of behavioral skills (e.g. breathing, relaxation, activity pacing, distraction, and calming statements). Participants also receive a specialized type of neuromuscular exercise training which focuses on core strength, gait and balance.
  Interventions: Behavioral: Fibromyalgia Integrative Training for Teens
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy (CBT) is a psychological coping skills training using education on gate control theory of pain, behavioral strategies such as muscle relaxation and activity pacing, and cognitive strategies including distraction, problem-solving, and using calming self-statements.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Graded Aerobic Exercise (Active Comparator): Graded aerobic exercise (GAE) utilizes a circuit-training approach with short intervals of exercise interspersed with brief rest breaks.
  Interventions: Behavioral: Graded Aerobic Exercise

INTERVENTIONS:
Behavioral: Fibromyalgia Integrative Training for Teens — This intervention will consist of 16 in-person group-based sessions held twice per week over 8 weeks. Sessions last 90 minutes and will be led jointly by a psychologist/therapist and exercise trainer using manualized protocols.
  Other Names: FIT Teens
  Arms: Fibromyalgia Integrative Training for Teens
Behavioral: Cognitive Behavioral Therapy — This intervention will consist of 16 in-person group-based sessions held twice per week over 8 weeks. Sessions last 90 minutes and will be led jointly by a psychologist/therapist and exercise trainer using manualized protocols.
  Other Names: CBT; coping skills
  Arms: Cognitive Behavioral Therapy
Behavioral: Graded Aerobic Exercise — This intervention will consist of 16 in-person group-based sessions held twice per week over 8 weeks. Sessions last 90 minutes and will be led jointly by a psychologist/therapist and exercise trainer using manualized protocols.
  Other Names: GAE
  Arms: Graded Aerobic Exercise

SUMMARY:
This study evaluated whether Fibromyalgia Integrative Training program for Teens (FIT Teens), a combined cognitive behavioral therapy and neuromuscular exercise training program is more effective in reducing disability in adolescents with Juvenile Fibromyalgia compared to cognitive behavioral therapy (CBT) alone or a graded aerobic exercise (GAE) program alone. One third of participants received the FIT Teens training; one third received CBT training; and one third of participants received the GAE training.

DETAILED DESCRIPTION:
Juvenile-onset fibromyalgia (JFM) is a chronic, debilitating pain condition that typically persists into adulthood for the majority of patients. Whereas medications offer limited and short-term symptom relief for JFM, our research group has demonstrated that cognitive-behavioral therapy (CBT) is safe, effective and durable in reducing functional disability and depressive symptoms in adolescents with this condition. However, 60% of patients receiving CBT did not show clinically significant improvement in functional disability, and pain levels remained in the moderate range despite being reduced overall. Our multidisciplinary team of experts in Behavioral Medicine, Rheumatology and Exercise Science has developed and tested the feasibility of a new Fibromyalgia Integrative Training program for Teens (FIT Teens), which enhances the established CBT intervention with a novel neuromuscular exercise training program derived from evidence-based pediatric injury prevention research. Pilot testing showed excellent patient engagement, no adverse effects and very promising early results indicating this treatment to have even stronger effects on disability and pain outcomes than CBT alone. This trial evaluated whether the FIT Teens intervention is more effective than CBT alone or graded aerobic exercise alone and whether treatment effects are sustainable over 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile Fibromyalgia diagnosis by pediatric rheumatologist or pain physician and confirmed by 2010 American College of Rheumatology (ACR) criteria modified for pediatric use
* Functional Disability Score ≥ 13, indicating at least moderate disability
* Average pain intensity in the past week ≥ 4 on a 0 -10 cm Visual Analog Scale
* Stable medications prior to enrollment

Exclusion Criteria:

* Comorbid rheumatic disease (e.g. juvenile arthritis, systemic lupus erythematous)
* Untreated major psychiatric diagnoses (e.g. bipolar disorder, psychoses, symptoms of major depression) or documented developmental delay
* Any medical condition determined by their physician to be a contraindication for physical exercise
* Taking opioid pain medication

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 389 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Kashikar-Zuck, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (7):
- United States (6):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Riley Children's Hospital-University of Indiana, Indianapolis, Indiana
  - Boston Chilldren's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kashikar-Zuck S, Briggs MS, Bout-Tabaku S, Connelly M, Daffin M, Guite J, Ittenbach R, Logan DE, Lynch-Jordan AM, Myer GD, Ounpuu S, Peugh J, Schikler K, Sugimoto D, Stinson JN, Ting TV, Thomas S, Williams SE, Zempsky W; Childhood Arthritis and Rheumatology Research Alliance (CARRA) Pain Workgroup Investigators. Randomized clinical trial of Fibromyalgia Integrative Training (FIT teens) for adolescents with juvenile fibromyalgia - Study design and protocol. Contemp Clin Trials. 2021 Apr;103:106321. doi: 10.1016/j.cct.2021.106321. Epub 2021 Feb 20. PMID 33618033
- [Background] Kashikar-Zuck S, Barnett KA, Williams SE, Pfeiffer M, Thomas S, Beasley K, Chamberlin LA, Mundo K, Ittenbach RF, Peugh J, Gibler RC, Lynch-Jordan A, Ting TV, Gadd B, Taylor J, Goldstein-Leever A, Connelly M, Logan DE, Williams A, Wakefield EO, Myer GD; FIT Teens Clinical Trial Study Group and the Childhood Arthritis and Rheumatology Research Alliance (CARRA) Pain Workgroup Investigators. FIT Teens RCT for juvenile fibromyalgia: Protocol adaptations in response to the COVID 19 pandemic. Contemp Clin Trials Commun. 2022 Nov 29;30:101039. doi: 10.1016/j.conctc.2022.101039. eCollection 2022 Dec. PMID 36467389
- [Derived] Kashikar-Zuck S, Thomas S, Bonnette S, Gibler RC, DiCesare C, Schille A, Hulburt T, Briggs MS, Ounpuu S, Myer GD; FIT Teens Clinical Trial Study Group. Comparison of Pain Characteristics, Strength, and Movement Patterns in Adolescents With Juvenile Fibromyalgia and High Versus Low Fear of Movement. J Pain. 2024 Sep;25(9):104586. doi: 10.1016/j.jpain.2024.104586. Epub 2024 May 31. PMID 38823603
- [Derived] Lynch-Jordan AM, Connelly M, Guite JW, King C, Goldstein-Leever A, Logan DE, Nelson S, Stinson JN, Ting TV, Wakefield EO, Williams AE, Williams SE, Kashikar-Zuck S; Fibromyalgia Integrative Training for Teens Clinical Trial Study Group and the Childhood Arthritis and Rheumatology Research Alliance Pain Workgroup Investigators. Clinical Characterization of Juvenile Fibromyalgia in a Multicenter Cohort of Adolescents Enrolled in a Randomized Clinical Trial. Arthritis Care Res (Hoboken). 2023 Aug;75(8):1795-1803. doi: 10.1002/acr.25077. Epub 2023 Feb 16. PMID 36537193

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the group-based nature of the study, potential participants completed their baseline (T1) assessment and then waited up to 4 weeks before treatment assignment. A potential participant would be excluded from the study prior to treatment assignment for the reasons of screen-fails, no longer interested in the study, starting a disallowed treatment, or are lost to contact.
Groups:
- Fibromyalgia Integrative Training for Teens: Fibromyalgia Integrative Training for Teens (FIT Teens) is a combined cognitive behavioral therapy and neuromuscular training.
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy (CBT) is a psychological pain coping skills training program.
- Graded Aerobic Exercise: Graded aerobic exercise (GAE) is a circuit-training exercise program with short intervals of aerobic exercise interspersed with brief rest breaks.
Period: Overall Study
Arm/Group | Fibromyalgia Integrative Training for Teens | Cognitive Behavioral Therapy | Graded Aerobic Exercise
Started | 103 | 110 | 104
Completed Primary Endpoint | 87 | 93 | 79
Completed (Completed Study) | 83 | 89 | 72
Not Completed | 20 | 21 | 32

BASELINE CHARACTERISTICS:
Population: While 389 participants were enrolled (signed consent and completed a pre-treatment assessment), 317 participants were randomized. This difference is due to screen-fails as well as those who voluntarily withdrew or were lost-to-contact prior to treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibromyalgia Integrative Training for Teens | Cognitive Behavioral Therapy | Graded Aerobic Exercise | Total
Number analyzed (Participants) | 103 | 110 | 104 | 317
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 103 | 110 | 104 | 317
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.73 (1.49) | 15.61 (1.61) | 15.96 (1.47) | 15.76 (1.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 97 | 99 | 294
  Male | 5 | 13 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 9 | 25
  Not Hispanic or Latino | 98 | 99 | 95 | 292
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 1 | 0 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 7 | 7 | 4 | 18
  White | 85 | 92 | 90 | 267
  More than one race | 8 | 8 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 3 | 0 | 3
  United States | 103 | 107 | 104 | 314
Functional Disability Inventory (FDI) [Mean (Standard Deviation); unit: units on a scale] — Functional Disability Inventory (FDI) is a 15-item self-report measure, developed to assess perceived difficulty in the performance of daily activities in home, school, recreational, and social domains due to pain. Total sum scores are calculated and range from 0 - 60, with higher scores indicating greater functional disability. Clinical reference points are: No/Minimal disability (0 to 12), Mild disability (13 to 20), Moderate disability (21 to 29) and Severe disability (≥30).
  units on a scale | 25.73 (8.67) | 24.05 (7.95) | 25.95 (8.33) | 25.22 (5.84)
Pain Intensity (VAS) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was measured using the Visual Analog Scale (VAS), which is a validated measure of pain intensity in children and adolescents. Participants were shown a line with the written anchors of "no pain" and "pain as bad as I can imagine" on either end.
  The line represents a 0-10 scale, where higher scores are representative of higher pain intensity with a score of 4-6 indicating at least moderate pain levels and a score of 7-10 indicating severe pain levels.
  units on a scale | 5.71 (1.30) | 5.93 (1.34) | 5.88 (1.26) | 5.84 (1.30)

OUTCOME MEASURES:

1. Primary Outcome: Functional Disability Inventory
Description: Functional Disability Inventory (FDI) is a validated 15-item self-report measure, developed to assess perceived difficulty in the performance of daily activities in home, school, recreational, and social domains due to pain. Total sum scores are calculated and range from 0 - 60, with higher scores indicating greater functional disability. Clinical reference points are: No/Minimal disability (0 to 12), Mild disability (13 to 20), Moderate disability (21 to 29) and Severe disability (≥30). For this primary outcome, data from this questionnaire was used to compare baseline response to 3 month follow up to examine whether a reduction in disability occurs.
  The main outcome measure for this comparison is the difference in baseline and primary endpoint (3 month) FDI scores for each of the three interventions (FIT Teens, CBT, and GAE).
Time Frame: Baseline to 3 month follow up (primary endpoint) and 6, 9 and 12 month follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fibromyalgia Integrative Training for Teens | Cognitive Behavioral Therapy | Graded Aerobic Exercise
Number analyzed (Participants) | 103 | 110 | 104
score on a scale
  Baseline | 25.78 [24.08 to 27.48] | 24.10 [22.31 to 25.89] | 25.96 [23.88 to 28.03]
  3-month endpoint | 21.83 [20.19 to 23.48] | 21.65 [19.86 to 23.43] | 24.70 [22.60 to 26.80]
  6-month endpoint | 21.26 [19.49 to 23.02] | 21.01 [19.09 to 22.93] | 23.34 [20.88 to 25.80]
  9-month endpoint | 21.56 [19.46 to 23.66] | 20.71 [18.54 to 22.88] | 23.37 [20.82 to 25.92]
  12-month endpoint | 21.02 [18.71 to 23.33] | 20.15 [18.08 to 22.21] | 21.22 [18.56 to 23.87]

2. Secondary Outcome: Pain Intenstiy
Description: Pain intensity was measured using the Visual Analog Scale (VAS), which is a validated measure of pain intensity in children and adolescents. Participants were shown a line with the written anchors of "no pain" and "pain as bad as I can imagine" on either end.
  The line represents a 0-10 scale, where higher scores are representative of higher pain intensity with a score of 4-6 indicating at least moderate pain levels and a score of 7-10 indicating severe pain levels.
  This measure was completed daily for one week and scores averaged over that time. For this secondary outcome, data from this measure were used to compare baseline response to 3 month follow up to examine whether a reduction in pain intensity occurred.
Time Frame: Baseline to 3 month follow up (primary endpoint) and 6, 9 and 12 month follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fibromyalgia Integrative Training for Teens | Cognitive Behavioral Therapy | Graded Aerobic Exercise
Number analyzed (Participants) | 103 | 110 | 104
units on a scale
  Baseline | 5.71 [5.48 to 5.94] | 5.93 [5.66 to 6.21] | 5.88 [5.58 to 6.18]
  3-month endpoint | 5.29 [4.78 to 5.79] | 5.41 [4.95 to 5.87] | 5.44 [4.98 to 5.91]
  6-month endpoint | 5.27 [4.80 to 5.74] | 5.19 [4.76 to 5.62] | 5.42 [4.90 to 5.94]
  9-month endpoint | 5.07 [4.64 to 5.50] | 5.13 [4.73 to 5.54] | 5.45 [4.92 to 5.98]
  12-month endpoint | 4.91 [4.46 to 5.35] | 4.88 [4.48 to 5.28] | 5.18 [4.70 to 5.66]

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning at time of consent through the final endpoint (12-months post treatment end), approximately 14 months total.
Description: General clinicaltrials.gov definitions apply; however, body systems vary to align with common AEs reported in this population. Our systematic approach for the assessment of AEs included asking participants about changes in their health at each assessment visit. Coordinators also received alerts through EMRs when participants were in the ER. Additionally, AEs could be spontaneously reported during treatment sessions. AEs considered possibly, likely or definitely related are reported here.
Arm/Group | Fibromyalgia Integrative Training for Teens | Cognitive Behavioral Therapy | Graded Aerobic Exercise
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/110 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/110 | 0/104
Other Adverse Events (participants affected / at risk) | 12/103 | 10/110 | 16/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibromyalgia Integrative Training for Teens (N=103) | Cognitive Behavioral Therapy (N=110) | Graded Aerobic Exercise (N=104)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia/palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Extremity pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 9 (9)
Generalized weakness/pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Sprain/strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Heat syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Increased emotional distress (Psychiatric disorders) | 4 (4) | 3 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT03268421/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT03268421/SAP_001.pdf